CLINICAL TRIAL: NCT01275976
Title: Effect of C1-esterase Inhibitor on Systemic Inflammation in Trauma Patients With a Femur or Pelvic Fracture
Acronym: CAESAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility and limited feasibility
Sponsor: UMC Utrecht (Other)
Collaborators: Prothya Biosolutions (Industry)
Responsible Party: Principal Investigator, Prof. dr Leenen, L.P.H. Leenen, MD, PhD, UMC Utrecht., UMC Utrecht
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 34932
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Trauma; Inflammation; Sepsis; Multiple Organ Dysfunction Syndrome
Keywords: C1-esterase inhibitor; Systemic inflammation; Sepsis; Trauma; Multiple Organ Dysfunction Syndrome; Cytokines
MeSH Terms: conditions — Wounds and Injuries; Inflammation; Sepsis; Multiple Organ Failure; Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C1-esterase inhibitor (Active Comparator): C1-esterase inhibitor, 100 U/kg bodyweight
  Interventions: Drug: C1-esterase inhibitor
- Saline 0.9% (Placebo Comparator): Saline 0.9%
  Interventions: Other: Saline 0.9%

INTERVENTIONS:
Drug: C1-esterase inhibitor — C1-esterase inhibitor 200 U/kg infusion over 30 minutes, just before the start of the femur or pelvic fixation operation.
  Other Names: Cetor® (RVG 19303)
  Arms: C1-esterase inhibitor
Other: Saline 0.9% — Infusion, just before the start of the femur or pelvic fixation operation
  Arms: Saline 0.9%

SUMMARY:
Trauma and major operation are associated with an excessive inflammation reaction due to tissue injury. This overwhelming immune response is considered to be a major risk factor in the pathogenesis of late inflammatory complications such as acute respiratory distress syndrome (ARDS), multiple organ dysfunction syndrome (MODS) and sepsis.

The investigators hypothesize that administration of C1-esterase inhibitor (C1-INH) will attenuate the humane inflammatory response and, thereby, reduce the risk of inflammatory complications due to surgical interventions in trauma patients with a femur or pelvic fracture

DETAILED DESCRIPTION:
Systemic inflammation in response to a femur or pelvic fracture and fixation is associated with complications, such as acute respiratory distress syndrome (ARDS) and multiple organ dysfunction syndrome (MODS). The injury itself, but also the additional fixation procedure give a release of pro-inflammatory cytokines, in particular interleukin (IL)-6. This results in an aggravation of the initial systemic inflammatory response, and will cause in some patients an increased risk on the development of inflammatory complications, like ARDS and MODS. Which can lead to higher morbidity, mortality and prolonged hospital stay.

Various strategies, such as damage control orthopedics, have been proposed to prevent these complications. Another strategy is to decrease the inflammatory reaction caused by the surgical procedure, and by interventions focused on inhibition of the innate inflammatory response. This will lower the risk of complications.

A promising candidate is the endogenously produced serum protein C1-esterase inhibitor (C1-INH). This protein is an acute phase protein, produced by the liver in response to inflammatory conditions. C1-INH is a major inactivator of the complement system, but important additional anti-inflammatory properties have been demonstrated. A previous study of from our laboratory showed that administration of the drug C1-INH significantly reduced the concentration of circulating pro-inflammatory cytokines such as IL-6, during human experimental endotoxemia. Treatment with C1-INH has been proven to be safe in treatment with humans, even in high dosages and in pregnant patients with C1-INH deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Multi trauma patients
* Femur or pelvic fracture
* Injury Severity Score (ISS) ≥ 18
* Age 18-80 yrs

Exclusion Criteria:

* Congenital C1-inhibitor deficiency
* Use of immune suppressants
* Pregnancy
* Known hypersensitivity for blood products
* Fixation of femur fracture with external fixation or osteosynthesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Delta Interleukine-6 | 6 hours after C1-INH administration

SECONDARY OUTCOMES:
Cytokines and other markers of inflammation | up to 12 days after C1-INH administration
Neutrophil redistribution and phenotype | Up to 12 days after C1-INH administration
C1-inhibitor and complement concentration and activity | Up to 12 days after C1-INH administration
Hemodynamic response | Up to 12 days after C1-INH administration

CONTACTS AND LOCATIONS:
Overall Officials: Luke P Leenen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Centre Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Heeres M, Visser T, van Wessem KJ, Koenderman AH, Strengers PF, Koenderman L, Leenen LP. The effect of C1-esterase inhibitor on systemic inflammation in trauma patients with a femur fracture - The CAESAR study: study protocol for a randomized controlled trial. Trials. 2011 Oct 11;12:223. doi: 10.1186/1745-6215-12-223. PMID 21988742